CLINICAL TRIAL: NCT00019344
Title: A Phase I Trial of Daily Bolus Flavopiridol for Five Consecutive Days in Patients With Refractory Neoplasms
Brief Title: Flavopiridol in Treating Patients With Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065779; NCI-97-C-0171C; NCI-T97-0064; NCT00001585 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2004-04-21 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2002-05

CONDITIONS: Lymphoma; Prostate Cancer; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; stage IV prostate cancer; recurrent prostate cancer; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Prostatic Neoplasms; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — alvocidib

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of flavopiridol in treating patients who have refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose-limiting toxicity and maximum tolerated dose of flavopiridol in patients with refractory solid tumors or lymphoma. 2. Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients receive flavopiridol IV over 1 hour on day 1. Treatment continues every 3 weeks in the absence of disease progression. A cohort of 3-6 patients receives treatment at each dose level of flavopiridol. If dose-limiting toxicity (DLT) occurs in no more than 1 of 6 patients, subsequent cohorts of 6 patients each receive escalating doses of drug on the same schedule. Intrapatient dose escalation to the next level is permitted in the absence of DLT.

PROJECTED ACCRUAL: Approximately 36 patients will be accrued for this study within 27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven refractory solid tumor or lymphoma requiring systemic therapy No standard therapeutic options exist Prostate cancer patients: Tumor progression during blockade of testicular and adrenal androgen required PSA elevation on 2 consecutive blood samples, 2 weeks apart Serum testosterone concentrations in the castrate range Leuprolide or other gonadotropin-releasing hormone (GnRH) analogs maintained if no prior orchiectomy No CNS neoplasms

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count at least 75,000/mm3 Absolute granulocyte count at least 1,000/mm3 No active coagulopathy requiring therapeutic anticoagulation Hepatic: SGOT and SGPT no greater than 2.5 times normal Bilirubin no greater than 1.5 times normal (3 times normal if Gilbert's disease present) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of unstable or newly diagnosed angina pectoris No myocardial infarction within past 6 months No New York Heart Association class II-IV heart disease Other: No serious concurrent medical illness HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No prior flavopiridol Endocrine therapy: See Disease Characteristics A least 4 weeks since prior flutamide or other antiandrogen therapy without disease improvement At least 4 weeks since prior hormonal therapy for breast carcinoma and must show evidence of disease progression No concurrent corticosteroids except for physiological replacement Radiotherapy: At least 4 weeks since prior radiotherapy and recovered At least 6 weeks since prior bone-seeking radioisotope therapy Surgery: Not specified Other: At least 3 months since prior suramin treatment At least 2 months since prior UCN-01 No concurrent anticoagulation therapy No other concurrent antineoplastic therapy except for GnRH for prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-08

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Sausville, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States

REFERENCES:
- [Result] Senderowicz AM, Messmann R, Arbuck S, et al.: A phase I trial of 1 hour infusion of flavopiridol (FLA), a novel cyclin-dependent Kinase inhibitor, in patients with advanced neoplasms. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-796, 2000.